CLINICAL TRIAL: NCT06105697
Title: Effect of Aerobic Blood Flow Restriction Training in Academy Football Players: A Randomised Controlled Trial
Brief Title: Effects of Aerobic Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 361CER23
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2023-11

CONDITIONS: Aerobic Exercise; Blood Flow Restriction Therapy
Keywords: Blood Flow Restriction; Aerobic Capacity; Soccer; Repeat Sprint Ability; Countermovement Jump

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction (Experimental I) (Experimental): Running with Blood Flow Restriction on the treadmill for 4 sets of 5 minutes,1' interset rest using a periodization methodology in soccer (Match Day 4 and Match Day 3).
  Interventions: Other: Blood flow restriction Running on Treadmill
- Non-Blood flow restriction (Experimental II) (Experimental): Running without Blood Flow Restriction on the treadmill for 4 sets of 5 minutes,1' interset rest using a periodization methodology in soccer (Match Day 4 and Match Day 3).
  Interventions: Other: Running on Treadmill

INTERVENTIONS:
Other: Blood flow restriction Running on Treadmill — Soccer players included in experimental group I will carry out this program for 6 weeks, setting the blood pressure to ~ 60% of limb occlusion pressure (AOP). They will run for 4 sets of 5 minutes, separated by 1 minute of rest, at 50-60% of their maximum Aerobic Speed.
  Arms: Blood flow restriction (Experimental I)
Other: Running on Treadmill — Soccer players included in experimental group II will carry out the program for 6 weeks without occlude the blood pressure. They will run for 4 sets of 5 minutes, separated by 1 minute of rest, at 50-60% of their maximum Aerobic Speed.
  Arms: Non-Blood flow restriction (Experimental II)

SUMMARY:
The aim is to evaluate the effects of aerobic blood flow restriction on academy football players. Randomized clinical trial, with two intervention groups: Experimental group I will carry out training based on running on the treadmill using blood flow restriction (BFR) on match days 4 and 3 pre-competition (MD-4, MD-3). On the other hand, the Experimental II group will perform the same training without the use of BFR for 6 weeks. The study will be carried out during the 2023-2024 season in the National and Youth Honor Divisions of Spanish soccer, with soccer teams from Mallorca Island. Before and after 6 weeks of intervention, the countermovement jump (CMJ), maximum aerobic speed (MAS), VO2max, and repeat sprint ability will be evaluated. The levels of muscle soreness (DOMS) will be evaluated at MD-4, MD-3, and MD-2. The same procedure will be carried out to evaluate muscle fatigue, sleep quality, and stress through a questionnaire. Sociodemographic and anthropometric data will be collected before starting the study. In addition, the rate of exertion perceived will be evaluated at MD-4, MD-3, and MD-2.

DETAILED DESCRIPTION:
The warm-up will consist of federation Internationale football association (FIFA) 11+. In addition, the warm-up will contain a familiarization with the jump test.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* No injuries players

Ages: 15 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Countermovement Jump (CMJ) | Change from Baseline in countermovement Jump (CMJ Test) at 6 weeks
  CMJ Test measured by Force Platform (Vald Performance, Brisbane, Australia)
Change from Baseline in Treadmill Incremental Test | Change from Baseline in Maximum Aerobic Speed at 6 Weeks
  Maximum Aerobic Speed (MAS) measured by the Treadmill Incremental test
Change from Baseline in Repeat Sprint Ability | Change from Baseline in Repeat Sprint Ability at 6 Weeks
  Repeat Sprint Ability measured by the Bangsbo Test
Change from Baseline In Yoyo Intermittent Recovery Test Level 1 | Change from Baseline in Yoyo Intermittent Recovery Level 1 at 6 Weeks
  Vo2max Indirect measured by the Yoyo Intermittent Recovery Test Level I

SECONDARY OUTCOMES:
Change from Baseline in Rating of Perceived Exertion (RPE) | Change from Baseline in RPE at Match Day -4 (MD-4), MD-3, MD-2 during the 6 Weeks´ Intervention
  Rating of Perceived Exertion (RPE) measured by Borg scale (0=Rest; 1=Really easy; 2=easy; 3=moderate; 4=sort of hard; 5=hard; 6=hard; 7=Really hard; 8= Really hard; 9= Really, really, hard; 10= Maximal)
Change from Baseline in Fatigue | Change from Baseline in Fatigue at Match Day -4 (MD-4), MD-3, MD-2 during the 6 Weeks´ Intervention
  Fatigue measured by a Wellness Questionary (1= Always tired; 2=More tired than normal; 3=Normal; 4= Fresh; 5= Very fresh)
Change from Baseline in Muscle Soreness | Change from Baseline in Muscle Soreness at Match Day -4 (MD-4), MD-3, MD-2 during the 6 Weeks´ Intervention
  Muscle Soreness measured by a Wellness Questionary (1=Very sore; 2= Increase in soreness/ tightness; 3=Normal; 4=Feeling good; 5=Feeling great)
Change from Baseline in Sleep Quality | Change from Baseline in Sleep Quality at Match Day -4 (MD-4), MD-3, MD-2 during the 6 Weeks´ Intervention
  Sleep Quality measured by a Wellness Questionary (1=Insomnia; 2=Restless sleep; 3=Difficulty falling asleep; 4=good; 5=Very restful)
Change from Baseline in Stress | Change from Baseline in Stress at Match Day -4 (MD-4), MD-3, MD-2 during the 6 Weeks´ Intervention
  Stress measured by a Wellness Questionary (1=Highly stressed; 2=Feeling stressed; 3=Normal; 4=Relaxed; 5=Very relaxed)
Change from Baseline in Mood | Change from Baseline in Stress at Match Day -4 (MD-4), MD-3, MD-2 during the 6 Weeks´ Intervention
  Mood measured by a Wellness Questionary (1=Highly annoyed / irritable / down; 2=Snappy with team-mates, family and friends; 3=Less interested in others / activities; 4=Generally good mood; 5=Very positive mood)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero Franco, PhD, Study Director — University of the Balearic Islands; Christian Castilla López, MsC, Principal Investigator — University of the Balearic Islands
Locations (2):
- Spain (2):
  - Christian, Palma de Mallorca, Balearic Islands
  - University of the Balearic Islands, Palma de Mallorca, Balearic Islands

IPD SHARING:
Plan to Share IPD: No